CLINICAL TRIAL: NCT02291159
Title: Effectiveness of Dry Needling (DNHS Technique) in the Treatment of Upper Limb Spasticity and Function in Stroke Patients: a Randomized Clinical Trial
Brief Title: Effects of DNHS Technique in the Treatment of Upper Limb Spasticity and Function in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Pablo Herrero Gallego, Dr. Pablo Herrero Gallego, Universidad San Jorge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USJ_DNHS_UL_01
Record Dates: First submitted 2014-11-10; First posted 2014-11-14 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Stroke; Spasticity
Keywords: stroke; spasticity; dry needling; upper motor neuron syndrome; motor function
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention-DNHS technique (Experimental): Dry needling of Myofascial Trigger Points
  Interventions: Device: DNHS ® (Dry Needling for Hypertonia and Spasticity)
- Control-Sham Dry Needling (Sham Comparator): Sham Dry Needling of Myofascial Trigger Points
  Interventions: Device: Sham Dry Needling

INTERVENTIONS:
Device: DNHS ® (Dry Needling for Hypertonia and Spasticity) — Dry needling of Myofascial Trigger Points. 2 sessions, one per week, in biceps brachii, brachialis, flexor digitorum superficialis nad profundus, adductor pollicis and first dorsal interossei
  Arms: Intervention-DNHS technique
Device: Sham Dry Needling — Sham dry needling of Myofascial Trigger Points. 2 sessions, one per week, in biceps brachii, brachialis, flexor digitorum superficialis nad profundus, adductor pollicis and first dorsal interossei
  Arms: Control-Sham Dry Needling

SUMMARY:
Introduction: Stroke is a neurological deficit caused by a decrease in cerebral blood flow. The DNHS ® (Dry Needling for hypertonia and Spasticity) technique is a dry needling technique to reduce spasticity and hypertonia and improve function in patients with CNS injury. The main objective of this trial is to analyze the therapeutic effect of DNHS® technique in motor function in patients between 45 and 80 in a chronic state after a stroke. Methods: Double-blinded randomized clinical trial. There will be an intervention group (DNHS® technique) and a sham control group. The intervention will be 2 sessions, one per week, in biceps brachii, brachialis, flexor digitorum superficialis nad profundus, adductor pollicis and first dorsal interossei. The Fugl Meyer Assessment Scale, Modified Ashworth Scale and Stroke Impact Scale will be used as outcome measures. The data will be expressed as mean ± (Standard Deviation). The standardized difference or effect size (ES, 90% confidence limit) in the selected variables will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* people aged 40-85 years with hemiplegia resulting from stroke of more than 6 months evolution (chronic stroke)
* ability to follow instructions and reply to assessment questonnaires

Exclusion Criteria:

* recurrent stroke episodes
* other concomitant neurodegenerative conditions
* fear to needles
* participation in a parallel study
* any absolute contraindication for deep dry needling

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment Scale (Motor Function) | Two weeks

SECONDARY OUTCOMES:
Modified Ashworth Scale (Hypertonia/Spasticity) | Two weeks
Impact Stroke Scale (Quality of Life) | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Herrero Pablo, Dr., Study Director — San Jorge University
Locations (1):
- San Jorge University, Villanueva de Gállego, Zaragoza, Spain